CLINICAL TRIAL: NCT02176057
Title: Nepal Elimination of Trachoma Study
Acronym: NETS
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Nepal Ministry of Health implemented public drug treatment prior to the proposed start date
Sponsor: University of California, San Francisco (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NETS-13-10961; K23EY019881 (NIH)
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Trachoma
Keywords: trachoma
MeSH Terms: conditions — Trachoma | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Antibiotic (Experimental): Azithromycin, suspension (liquid), 1 gram, one-time dose
  Interventions: Drug: Azithromycin
- Observation (No Intervention)

INTERVENTIONS:
Drug: Azithromycin
  Other Names: Zithromax
  Arms: Antibiotic

SUMMARY:
The main purpose of this study is to determine if ocular Chlamydia trachomatis infection can be eliminated in communities in Nepal following mass antibiotic distributions with azithromycin. The investigators will study both clinical trachoma and ocular C. trachomatis infection. The overall objective is to determine if the current World Health Organization (WHO) treatment strategy results in elimination of trachoma and infection.

1. The investigators hypothesize that 24 communities in Kanchanpur, Kailali, and Achham districts of Nepal which receive mass antibiotic treatments will achieve elimination of trachoma as a public health problem (clinical disease <5% in children 1-9 years old) more frequently than communities which have not received antibiotic treatments.
2. The investigators hypothesize that infection with C. trachomatis will be undetectable in all members within a community following mass treatment as determined by the most highly sensiti1. The investigators hypothesize that 24 communities in Kanchanpur, Kailali, and Achham districts of Nepal which receive mass antibiotic treatments will achieve elimination of trachoma as a public health problem (clinical disease <5% in children 1-9 years old) more frequently than communities which have not received antibiotic treatments.

2. The investigators hypothesize that infection with C. trachomatis will be undetectable in all members within a community following mass treatment as determined by the most highly sensitive nucleic acid amplification testing available (mRNA-based APTIMA and DNA-based AMPLICOR PCR).ve nucleic acid amplification testing available (mRNA-based APTIMA and DNA-based AMPLICOR PCR).

DETAILED DESCRIPTION:
Here we evaluate whether ocular chlamydia infection and clinical trachoma are eliminated from 24 communities in western Nepal following a mass antibiotic distribution program. It is unknown if repeated treatments should continue or can be stopped thereby minimizing side effects and the high cost of medicine distribution. The investigators plan to randomize individuals to two groups to study the effects of a mass antibiotic distribution program: 1) treatment of antibiotics and 2) delayed treatment of antibiotics (after 4-6 months).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-9 years
* Children who live in Kailai, Kanchanpur, or Achham Districts of Nepal

Exclusion Criteria:

* All individuals who are allergic to macrolides
* All pregnant woman
* All neonates

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Trachoma (clinical and C. trachomatis) | 12 months

SECONDARY OUTCOMES:
Anthropometry (height for weight) | 12 months
Malaria | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Gaynor, MD, Principal Investigator — UCSF F. I. Proctor Foundation (California, USA)
Locations (1):
- Geta Eye Hospital, Geṭā, Kailali, Nepal